CLINICAL TRIAL: NCT03771222
Title: Prophylactic Donor Lymphocyte Infusion After Allo-PBSCT for Patients With Very High-risk Hematologic Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Head of Hematology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pDLI2018
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Donor Lymphocyte Infusion; Peripheral Blood Stem Cell Transplantation; Relapse; Graft-versus-host Disease; Decitabine
MeSH Terms: conditions — Recurrence; Graft vs Host Disease | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic DLI (Experimental): The scheduled time of the first prophylactic DLI was +30 ~ +60 days after transplantation for HLA-matched sibling donors (MSD)-PBSCT recipients and +60 ~ +90 days after transplantation for HLA-haploidentical sibling donors (HID)-PBSCT recipients.
  Interventions: Biological: Prophylactic DLI
- No prophylactic DLI (No Intervention)

INTERVENTIONS:
Biological: Prophylactic DLI — The G-CSF-mobilized PBSCs from cryopreserved cells of the graft were infused to the recipient at a dose of 2X10^7 CD3+ cells/kg recipient body weight. Decitabine (10 mg/m2, days 1 to 5) followed by prophylactic DLI would be given to those patients carrying TET2, DNMT3a or TP53 gene mutations.
  Other Names: Decitabine (trade name Dacogen)
  Arms: Prophylactic DLI

SUMMARY:
Unmanipulated allogenic peripheral blood stem cell transplantation (allo-PBSCT) has been an established treatment to cure high-risk leukemia/lymphoma. Relapse is the main cause of treatment failure for patients with relapsed/refractory disease or with very high-risk gene mutations such as TP53, TET2 and DNMT3a. Donor lymphocyte infusion (DLI) is an option to reduce relapse after allo-PBSCT for very high-risk disease without effective targeted therapy. In this study, the investigators aimed to compare the safety and efficacy of prophylactic DLI with G-CSF-primed peripheral blood progenitors for prevention of relapse after allo-PBSCT in patients with very high-risk leukemia/lymphoma.

DETAILED DESCRIPTION:
Conventional DLI has invariably been associated with high rates of severe graft-versus-host disease (GVHD) and GVHD-related non-relapse mortality (NRM). Thus, in our previous studies, the DLI procedure has been modified to use G-CSF-mobilized peripheral blood stem cells (PBSCs) instead of steady-state lymphocytes. G-CSF mobilization results in the modulation of the polarization potential of T cells from Th1 to Th2. In addition, T-cell hyporesponsiveness is induced via the proliferation of dendritic cell 2 and monocytes and the down-regulation of CD28/B7. Furthermore, G-CSF augments NK-T-cell-dependent CD8+ cytotoxicity. These data constructed the rationale for the use of G-CSF-primed peripheral blood DLI to reduce DLI-associated GVHD and enhance the GVT effect of DLI. To date, there is no effective target therapy for acute leukemia with gene mutations such as DNMT3A, TET2 and TP53 and their response to chemotherapy and survival even after allogenic stem cell transplantation remains poor. Hypomethylating agents were reported to reverse the repression of HLA molecules and cancer testis antigens on leukemia cells, rendering them more sensitive to anti-leukemic activity mediated by DLI. The use of low-dose decitabine after allogenic stem cell transplantation was safe for early hematopoietic reconstitution. Therefore, decitabine was planned to be given prior to prophylactic DLI in the current study.

ELIGIBILITY:
Inclusion Criteria:

* disease in the non-remission (NR) state prior to transplantation, including primary induction failure, relapse untreated or refractory to reinduction chemotherapy.
* achieving CR1 with ≥3 cycles of induction of chemotherapy.
* carrying TP53, DNMT3a, TET2 or FLT3-ITD gene mutation.

Exclusion Criteria:

* early relapse, either molecular relapse or hematological relapse.
* primary or secondary graft failure.
* concomitant uncontrolled disease and/or organ dysfunction (infection, severe heart, renal, respiratory or hepatic failure…).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse at 1 year after randomization | 1 year
  Relapse was defined as hematologic recurrence of malignancies after transplantation. Cumulative incidence of relapse was analyzed in a competing risk framework using Gray's method.
Cumulative incidence of non-relapse mortality (NRM) at 1 year after randomization | 1 year
  NRM was deﬁned as death from any cause without relapse. Cumulative incidence of NRM was analyzed in a competing risk framework using Gray's method.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) at 1 year after randomization | 1 year
  RFS will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test. Survival will be calculated from the date of randomization.
Cumulative incidence of acute GVHD at 100 days after randomization | 100 days
  The cumulative incidence of acute GVHD was estimated considering the competing risks.
Cumulative incidence of chronic GVHD at 1 year after randomization | 1 year
  The cumulative incidence of chronic GVHD was estimated considering the competing risks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No